CLINICAL TRIAL: NCT01605149
Title: Type 1 DM Bone Mineral Density in Childhood and Adolescence
Brief Title: Type 1 Diabetes Mellitus Bone Mineral Density in Childhood and Adolescence
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Laura Armas, Assistant Professor, Creighton University
Other Study IDs: 12-16425
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Case: Patients with Type 1 Diabetes Mellitus

SUMMARY:
Type 1 Diabetes Mellitus is a disease that has an effect on bone mineral density. It is unclear how and when it effects the bone density. The investigators are studying the effects of diabetes on bone mass compared to children without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit children from age 5 to age 18 with a diagnosis of Type 1 DM. Children will have various lengths of time since diagnosis.

Exclusion Criteria:

* We will exclude children on anticonvulsants or steroids and children with other concomitant illnesses that interfere with bone mass accrual, except for hypothyroidism on treatment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with Type 1 DM
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura AG Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States